CLINICAL TRIAL: NCT02161731
Title: Effect of Evacetrapib on the Pharmacokinetics and Pharmacodynamics of Warfarin in Healthy Subjects
Brief Title: Study of Evacetrapib (LY2484595) and Warfarin in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 15366; I1V-MC-EIBN (Other: Eli Lilly and Company)
Record Dates: First submitted 2014-06-10; First posted 2014-06-12 (Estimated); Results first posted 2018-10-03 (Actual); Last update posted 2018-10-03 (Actual); Status verified 2018-02

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — evacetrapib; Warfarin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Warfarin (Active Comparator): 15 milligram (mg) warfarin administered as a single oral dose on Day 1
  Interventions: Drug: Warfarin
- Evacetrapib + Warfarin (Experimental): Evacetrapib administered once daily (QD), orally, for 16 days with 15 mg warfarin co-administered once orally on Day 17
  Interventions: Drug: Evacetrapib; Drug: Warfarin

INTERVENTIONS:
Drug: Evacetrapib — Oral administration
  Other Names: LY2484595
  Arms: Evacetrapib + Warfarin
Drug: Warfarin — Oral administration

SUMMARY:
All study participants will receive both warfarin and a study drug called evacetrapib. The main purpose of this study is to look at how much warfarin gets into the blood stream and how long it takes the body to get rid of warfarin when given both with and without evacetrapib. Another purpose is to evaluate the effectiveness of warfarin therapy to prevent blood clots when given with evacetrapib by measuring the time it takes for blood to clot and comparing it to an average of the international normalized ratio (INR). INR measures the time it takes for blood to clot and compares it to an average.

The study will last approximately 5 weeks, not including screening.

ELIGIBILITY:
Inclusion Criteria:

* Participants have given written informed consent approved by Lilly and the ethical review board (ERB) governing the site
* A medical history and physical examination consistent with a being a healthy individual
* Male participants will use a reliable method of birth control (as deemed by the investigator) and not donate sperm during the study and for 3 months following the last dose of the investigational product
* Female participants are not of child-bearing potential due to surgical sterilization (at least 6 weeks after surgical hysterectomy, bilateral oophorectomy, or tubal ligation) confirmed by medical history, or post-menopausal
* Have a body mass index of 18 to 32 kilograms per square meter (kg/m^2)
* Participants are predicted to be cytochrome P450 2C9 (CYP2C9) extensive metabolizers as determined by genotyping assessment

Exclusion Criteria:

* Have an abnormality in the 12-lead electrocardiogram (ECG) that increases the risks associated with participating in the study
* Have an abnormal supine blood pressure
* Have a history or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; of constituting a risk when taking the study medication; or of interfering with the interpretation of data
* Show evidence of human immunodeficiency virus (HIV) infection and/or positive human HIV antibodies
* Show evidence of hepatitis C and/or positive hepatitis C antibody or evidence of hepatitis B and/or positive hepatitis B surface antigen
* Women who are pregnant or are lactating
* Have used or intend to use over-the-counter or prescription medications (including vitamins/mineral supplements, herbal medicine) 14 days prior to enrollment and during the study
* Have consumed grapefruit, cranberries, or grapefruit- or cranberry-containing products within 7 days prior to the first dose of warfarin
* Have a history or presence of significant bleeding disorders that is, hematemesis, melena, severe or recurrent epistaxis, hemoptysis, clinically overt hematuria or intracranial hemorrhage, gastrointestinal ulcers with hemorrhage
* Have a personal or family history of coagulation or bleeding disorders or reasonable suspicion of vascular malformations, for example, cerebral hemorrhage, aneurysm or premature stroke (cerebrovascular accident less than 65 years of age)
* Have a history of major head trauma (with loss of consciousness) within the past year or minor head trauma (without loss of consciousness) within the last 3 months prior to screening or history of major surgery within 3 months of screening
* Have planned surgery within 14 days after the last day of dosing
* Have an international normalized ratio/prothrombin time (INR/PT), or activated partial thromboplastin time (aPTT) above the normal reference range or abnormal Protein S antigen and/or Protein C activity at screening

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2014-06; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Madison, Wisconsin, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Evacetrapib + Warfarin: Evacetrapib administered once daily (QD), orally, for 16 days on Days 7 - 22 with 15 mg warfarin co-administered once orally on Day 17.
Period: Period 1 (Day -1 to Day 7 Predose)
Arm/Group | Warfarin | Evacetrapib + Warfarin
Started | 24 | 0
Received 1 Dose of Study Drug | 24 | 0
Completed | 24 | 0
Not Completed | 0 | 0
Period: Period 2 (Day 7 Dosing to Day 23)
Arm/Group | Warfarin | Evacetrapib + Warfarin
Started | 0 | 24
Received 1 Dose of Study Drug | 0 | 24
Completed | 0 | 22
Not Completed | 0 | 2
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Warfarin Then Evacetrapib + Warfarin: 15 mg warfarin administered as a single oral dose on Day 1. Evacetrapib administered QD, orally, for 16 days, Days 7- 22 with 15 mg warfarin co-administered once orally on Day 17.
Arm/Group | Warfarin Then Evacetrapib + Warfarin
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.0 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 23
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 11
  White | 9
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve From Time Zero to Infinity (AUC[0-∞]) of S-Warfarin
Time Frame: Days 1 and 17: 0, 1, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120, and 144 hours following warfarin dose
Population: All participants who received a dose of study drug and had evaluable data for AUC [0-∞].
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour/milliliter (ng*h/mL)
Groups:
- Warfarin: 15 mg warfarin administered as a single oral dose on Day 1.
- Evacetrapib + Warfarin: Evacetrapib administered QD, orally, for 16 days, Days 7 - 22 with 15 mg warfarin co-administered once orally on Day 17.
Arm/Group | Warfarin | Evacetrapib + Warfarin
Number analyzed (Participants) | 24 | 23
nanogram*hour/milliliter (ng*h/mL) | 128 (23) | 114 (19)

2. Primary Outcome: PK: Maximum Observed Concentration (Cmax) of S-warfarin
Time Frame: Days 1 and 17: 0, 1, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120, and 144 hours following warfarin dose
Population: All participants who received a dose of study drug and had evaluable data for Cmax.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Warfarin | Evacetrapib + Warfarin
Number analyzed (Participants) | 24 | 23
nanograms per milliliter (ng/mL) | 4.20 (21) | 4.34 (29)

3. Secondary Outcome: PK: AUC[0-∞] of R-warfarin
Time Frame: Days 1 and 17: 0, 1, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120, and 144 hours following warfarin dose
Population: All participants who received a dose of study drug and had evaluable data for AUC[0-∞].
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Warfarin | Evacetrapib + Warfarin
Number analyzed (Participants) | 24 | 23
ng*h/mL | 287 (16) | 271 (17)

4. Secondary Outcome: PK: Cmax of R-warfarin
Time Frame: Days 1 and 17: 0, 1, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120, and 144 hours following warfarin dose
Population: All participants who received a dose of study drug and had evaluable data for Cmax of R- enantiomers of Warfarin.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Warfarin | Evacetrapib + Warfarin
Number analyzed (Participants) | 24 | 23
ng/mL | 5.03 (21) | 5.27 (27)

5. Secondary Outcome: Pharmacodynamics (PD): Area Under the International Normalized Ratio Curve (AUC[INR]) of Warfarin
Description: The INR is a standardized ratio of the prothrombin time (PT), time it takes for blood to clot. AUC[INR] is the time curve used to measure change in INR over time.
Time Frame: Days 1 and 17: 0, 1, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120, and 144 hours following warfarin dose
Population: All participants who received a dose of study drug and had evaluable data for AUC[INR].
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio times hour (ratio*h)
Arm/Group | Warfarin | Evacetrapib + Warfarin
Number analyzed (Participants) | 24 | 23
ratio times hour (ratio*h) | 174 (7.0) | 165 (5.0)

6. Secondary Outcome: PD: Maximum Observed International Normalized Ratio Response (INRmax) of Warfarin
Time Frame: Days 1 and 17: 0, 6, 12, 24, 36, 48, 72, 96, 120, and 144 hours following warfarin dose
Population: All participants who received a dose of study drug and had evaluable date for INRmax.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Warfarin | Evacetrapib + Warfarin
Number analyzed (Participants) | 24 | 23
ratio | 1.47 (18) | 1.34 (11)

ADVERSE EVENTS:
Groups:
- 15 mg Warfarin: 15 milligram (mg) warfarin administered as a single oral dose on Day 1.
- 130 mg Evacetrapib: 130 mg Evacetrapib administered once daily (QD), orally, for 16 days, Days 7 - 22.
- 15 mg Warfarin + 130 mg Evacetrapib: Evacetrapib administered once daily (QD), orally, for 16 days, Days 7 - 22 with 15 milligram (mg) warfarin co-administered once orally on Day 17.
Arm/Group | 15 mg Warfarin | 130 mg Evacetrapib | 15 mg Warfarin + 130 mg Evacetrapib
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24 | 0/23
Other Adverse Events (participants affected / at risk) | 0/24 | 2/24 | 0/23
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 15 mg Warfarin (N=24) | 130 mg Evacetrapib (N=24) | 15 mg Warfarin + 130 mg Evacetrapib (N=23)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days